CLINICAL TRIAL: NCT01584661
Title: The Continuity of Nutritional Care From the Hospital to the Community and Its Impact on Health and Functional Indicators Among Elderly Patients
Brief Title: The Continuity of Nutritional Care Among Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bait Balev Hospital (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Danit R Shahar, Prof, Ben-Gurion University of the Negev
Other Study IDs: ABB-1-2012
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Continuity of Nutritional Care; Health Care Use; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Compliance with nutritional care: The Inclusion criteria comprise patients who were treated nutritionally with food enrichment supplements during their hospitalization in "Bait Balev" and were discharged to their homes with dietary recommendations. Participants who are willing to participate will sign an informed consent form. For patients with cognitive impairment or dementia, as reported in their medical records, their formal primary caregiver or proxy will sign the informed consent form.
  Interventions: Behavioral: Dietary recommendations

INTERVENTIONS:
Behavioral: Dietary recommendations

SUMMARY:
Objectives:

1. To determine the level of compliance with nutritional recommendations (dietary and nutritional supplements) following discharge from hospitalization;
2. To identify barriers for post-discharge adherence to professional nutritional recommendations;
3. To determine the impact of adherence (high vs. low) to the nutritional treatment guidelines on functional and health indicators.

Working hypothesis:

High adherence to nutritional care after hospitalization will be associated with better functional and health outcomes.

DETAILED DESCRIPTION:
The proposed study will follow patients who were hospitalized in the rehabilitation departments at "Bait Balev". Patients who were treated with nutritional supplements by a dietitian during hospitalization and received dietary recommendations upon discharge will be followed for their adherence with the treatment recommendations. The impact of the level of adherence to the nutritional recommendations on health will be assessed.

C2. Experimental design:

This shall be a retrospective and prospective cohort study. Patients from the orthopedic and neurologic rehabilitation departments, who received nutritional intervention by nutritional supplements during hospitalization and were advised to receive nutritional enrichment at discharge, will be enrolled to the study. The main criteria for nutritional intervention during hospitalization and recommendation for supplements upon discharge include, among others, withdrawal of alternative nourishment, underweight, undernutrition, non-voluntary weight loss, low protein status and other criteria typical among this population during hospitalization. In order to assess the level of compliance with dietitian's recommendations upon discharge, only patients who were discharged to their homes will be followed. In order to increase the sample size, a retrospective cohort study will be conducted, in which patients from the same departments who were discharged in the last 3 months will be followed both retrospectively and prospectively.

Home visits will take place 3 and 6 months after discharge, during which the dietitian shall complete a questionnaire measuring the level of patient compliance to the nutritional recommendations, and in addition the patient or their legal guardian shall provide anamnesis in order to review the effect of compliance on health, functional, nutritional and social status (it should be noted that approx. 90% of the patients in the hospital belong to the Maccabi Health Care Services group, so the follow up of discharged patients in the community will be conducted with Maccabi Health Care Services).

ELIGIBILITY:
Inclusion Criteria:comprise patients who were treated nutritionally with food enrichment supplements during their hospitalization in "Bait Balev" and were discharged to their homes with dietary recommendations. Participants who are willing to participate will sign an informed consent form. For patients with cognitive impairment or dementia, as reported in their medical records, their formal primary caregiver or proxy will sign the informed consent form.

-

Exclusion Criteria:

* 1. Patients who were discharged to a Retirement home; 2. Palliative patients; 3. Patients who are not members of Maccabi Health Care Services. 4. Patients with enteral nutrition (PZ / PEG / PEJ)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study population Patients over the age of 65 who are members of Maccabi Health Care Services will be recruited for the current study. The Inclusion criteria comprise patients who were treated nutritionally with food enrichment supplements during their hospitalization in "Bait Balev" and were discharged to their homes with dietary recommendations. Participants who are willing to participate will sign an informed consent form. For patients with cognitive impairment or dementia, as reported in their medical records, their formal primary caregiver or proxy will sign the informed consent form.
Sampling Method: Non-Probability Sample
Dates: Start 2012-07; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Primary: Compliance with nutritional recommendations

SECONDARY OUTCOMES:
Health status

CONTACTS AND LOCATIONS:
Locations (1):
- Bait Balev, Bat Yam, Israel